CLINICAL TRIAL: NCT07242703
Title: Efficacy of Ultraviolet B Phototherapy in the Management of Resistant and Relapsing Tinea Corporis and Tinea Cruris
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hagar El Sayed, Dr Hagar El Sayed Abd El Ghani Anter, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NBUVB in resistant tinea
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Fungal Resistance
MeSH Terms: interventions — Itraconazole; Terbinafine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NBUVB (Experimental): Type of phototherapy
  Interventions: Device: NBUVB
- Medical treatment (Active Comparator): combined oral itraconazole and terbinafine.
  Interventions: Drug: Itraconazole + terbinafine

INTERVENTIONS:
Device: NBUVB — Phototherapy device
  Arms: NBUVB
Drug: Itraconazole + terbinafine — Antifungal drugs
  Arms: Medical treatment

SUMMARY:
This study aims to assess the efficacy of narrow-band ultraviolet B (NB-UVB) phototherapy as a standalone treatment in patients with resistant and recurrent tinea.

To evaluate the clinical and mycological improvement in response to NB-UVB therapy compared to standard anti-fungal treatment alone.

DETAILED DESCRIPTION:
Randomized, parallel-group, two-arm clinical trial. Arm A (NB-UVB group): Patients receive narrowband UVB phototherapy only.

Arm B (Itraconazole + Terbinafine group): Patients receive combined oral itraconazole and terbinafine.

Allocation will be 1:1 using concealed randomization.

Intervention:

Intervention (Arm A):

Patients in Arm A will receive narrowband UVB phototherapy (311 nm) three times per week for a total of 8 weeks.

Starting dose: 280-320 mJ/cm² (based on Fitzpatrick skin type)

Dose escalation: Increase by 10-20% each week as tolerated, with weekly monitoring for erythema or other adverse effects.

Follow-up: All Arm A patients will be re-evaluated clinically and mycologically 8 weeks after completing the 8-week NB-UVB course (i.e., at week 16 from baseline) to assess sustained response and relapse.

Intervention (Arm B):

Patients in Arm B will receive oral itraconazole plus terbinafine concurrently:

Itraconazole: 200 mg once daily for 8 weeks

Terbinafine: 250 mg once daily for 8 weeks

Follow-up: All Arm B patients will be re-evaluated clinically and mycologically 8 weeks after completing the 8-week antifungal course (also at week 16 from baseline) to assess sustained response and relapse.

Monitoring: Weekly observation for erythema or side effects.

A follow-up period of 8 weeks after the end of treatment will be included to assess relapse and sustained clinical/mycological improvement.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years.

Both sexes.

Clinical diagnosis of tinea corporis or cruris.

Failure of ≥4 weeks of systemic antifungal therapy (e.g., terbinafine or itraconazole).

No antifungal (topical or systemic) or corticosteroid treatment in the 2 weeks preceding enrollment.

Recurrent infection (≥2 relapses in the past 6 months)

Positive KOH microscopy and culture at baseline

Exclusion Criteria:

* Photosensitivity disorders or photosensitizing medications.

Xeroderma pigmentosa, LE or other photosensitive dermatoses. dermatomyositis.

Other skin conditions (psoriasis, eczema, etc.).

Known autoimmune diseases, immunosuppression, or coagulopathies..

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Dermatophytosis Severity Score (DSS) | 8 weeks